CLINICAL TRIAL: NCT02929667
Title: Abnormal Ventilatory Response to Carbon Dioxide: a Potential Biomarker for Seizure Induced Respiratory Depression & Modification by SSRI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rup Kamal Sainju (Other)
Responsible Party: Sponsor-Investigator, Rup Kamal Sainju, Clinical Assistant Professor of Neurology, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 201607761
Record Dates: First submitted 2016-07-26; First posted 2016-10-11 (Estimated); Results first posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Epilepsy; SUDEP
Keywords: Fluoxetine
MeSH Terms: conditions — Epilepsy; Sudden Unexpected Death in Epilepsy | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator): Subjects randomized to treatment arm will receive fluoxetine with titration schedule consisting of 10 mg per day for 1 week, 20 mg per day for 1 week, 40 mg per day for 2 weeks, 20 mg per day for 1 week and 10 mg per day for 1 week. Then stop.
  Interventions: Drug: Fluoxetine
- Control (Placebo Comparator): Subjects randomized to control arm will receive placebo with titration schedule consisting of 10 mg per day for 1 week, 20 mg per day for 1 week, 40 mg per day for 2 weeks, 20 mg per day for 1 week and 10 mg per day for 1 week. Then stop.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluoxetine — Standard 6 weeks titration, starting 10 mg per day.
  Other Names: Prozac
  Arms: Treatment
Drug: Placebo — Standard 6 weeks titration.
  Arms: Control

SUMMARY:
Sudden unexpected death in epilepsy patients (SUDEP) is devastating outcome for some patients with epilepsy. It ranks second only to stroke among neurological diseases in years of potential life lost. Patho-mechanisms of SUDEP remain not well understood, however peri-ictal respiratory dysfunction likely plays an important role in many cases.

Literature supports a critical role for the serotonergic system in central control of ventilation. Serotonin neurons in the raphe nuclei of the brainstem sense rising carbon dioxide and low pH, thereby stimulating breathing and arousal. These responses may serve as mechanisms that protect against asphyxia, particularly during sleep or the post-ictal state. In mouse models of seizure-induced sudden death, pre-treatment with selective serotonin reuptake inhibitor (SSRI) agents prevents death following seizures. Hence, the investigators hypothesize that a subset of drug resistant epilepsy patients who have impaired central chemo-responsiveness have a greater degree of peri-ictal respiratory depression, therefore a higher risk of SUDEP. The investigators further hypothesize that fluoxetine will improve central chemo-responsiveness and therefore will reduce peri-ictal respiratory depression.

DETAILED DESCRIPTION:
Sudden unexpected death in epilepsy (SUDEP) refers to the sudden, unexpected, nontraumatic, non-drowning, witnessed or unwitnessed death of an individual with epilepsy. Postmortem examination in such cases fails to reveal an obvious medical or toxicologic cause for the death, and patients who die from SUDEP are typically healthy apart from their epilepsy. The incidence of SUDEP in epilepsy patients is estimated to be 0.1 in 1000 patient years, and this rate increases to >9.3 per 1000 for those with durg resistant epilepsy (DRE) who are candidates for epilepsy surgery. Although thought to be rare, SUDEP is estimated to be responsible for 17% of all deaths in patients with epilepsy, and approximately 50% of all deaths in patients with DRE. It is second only to stroke among neurological diseases in YPLL because many who die of SUDEP are relatively young and therefore it is a major public health concern. While there are some acknowledged risk factors for SUDEP, the actual cause, or causes, of SUDEP is not known. Seizure induced respiratory depression is likely to be a major contributor in SUDEP in many cases.

Preliminary results from the ventilatory response to CO2 or hypercapnic ventilatory response (HCVR) study of patient with epilepsy in epilepsy monitoring unit (EMU) suggests prolonged period of CO2 elevation after seizures correlating with low HCVR. These findings suggest a defect in CO2 responsiveness in this high-risk population that may predispose to SUDEP. Serotonin nerve cells in the brain stem are responsible for detecting increases in CO2, and in response stimulating breathing and arousal from sleep. Fluoxetine is a selective serotonin reuptake inhibitor (SSRI) drug that increases availability of serotonin in the brain. As such, it may serve to stimulate breathing after seizures in patients with epilepsy who exhibit low CO2 sensitivity at baseline and this may alter SUDEP risk.

This study consists of a double blind randomized controlled clinical trial with a 6-week titration of an intervention. It is designed to evaluate primarily feasibility of a larger clinical trial testing efficacy of fluoxetine in modifying HCVR in patients with epilepsy while also collecting important secondary and exploratory outcomes that would be valuable for designing future larger studies.

We will evaluate challenges in screening, enrollment, randomization, and completion of study-related procedures by quantifying the numbers of subjects eligible for screening, the number of subjects enrolled in the study per month, the proportion of patients successfully completing the study, and the specific challenges at each step. We will also assess challenges in setting up and performing outpatient HCVR testing.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 18 or older
2. Patients with epilepsy
3. Native English speaker or adequate fluency in English to provide informed consent.
4. Female patients of child-bearing potential must be using an acceptable method of contraception, and willing to refrain from sexual intercourse during the study.

Exclusion Criteria:

1. Progressive neurological disease.
2. Clinical diagnosis of bipolar disease, panic disorder, psychosis or severe depression, or PHQ-9 score > 20
3. Patients with prior hospitalization related to depression or Electroconvulsive therapy.
4. History of suicidal ideation or intent in past or present
5. Clinical history or laboratory evidence of hepatic or renal insufficiency.
6. Pregnant or lactating women.
7. Current heavy alcohol use (>14 drinks per week for men or >7 drinks per week for women) or) known medical disorder related to alcohol use or current illicit drug use, other than marijuana and its derivatives.
8. Patients with recent use (<1 month) or already taking fluoxetine or other selective serotonin reuptake inhibitors (SSRIs).
9. Concurrent use of monoamine oxidase inhibitors, antipsychotic agents, antidepressant agents other than SSRIs or frequent use of triptan agents (>2/week).
10. History of a previous allergic reaction or adverse effects with fluoxetine, hypersensitive reaction-anaphylaxis; laryngeal edema; hives
11. History of serotonin syndrome.
12. History of uncontrolled pulmonary or cardiac illness.
13. Patients with hypercapnic ventilatory response (HCVR) slope of > 2.0
14. Patients with known prolong QT interval
15. Patients with family history of prolong QT interval
16. Patients with family history of sudden cardiac death under the age of 40 in a first degree relative.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rup Sainju, Principal Investigator — University of Iowa
Locations (2):
- United States (2):
  - The Univeristy of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Univeristy of Iowa Hospitals and Clinics, Iowa City, Iowa

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 30 subjects enrolled from February 2017 to February 2019. These 30 subjects underwent further screening before randomization to an intervention. Eight of the subjects failed to meet eligibility for randomization to an intervention, hence only 22 participants were randomized equally (1:1) to one of the treatment arms.
Pre-assignment Details: A total of 6 subjects with HCVR slope of > 2.0 L/min/mm Hg were excluded.Two additional subjects did not meet other inclusion criteria for randomization.
Period: Overall Study
Arm/Group | Treatment | Control
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 10 | 7 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Study Recruitment Rate
Description: Number of participants enrolled every 3 months.
Time Frame: From the date of enrollment every 3 months up to 2 years
Population: Due to being a feasibility study, recruitment is reported for the whole population (drug + placebo).
Measure: Mean (Full Range); unit: participants/3 months
Groups:
- Recruitment: Number of subjects (both fluoxetine and placebo arms) enrolled in the study.
Arm/Group | Recruitment
Number analyzed (Participants) | 30
participants/3 months | 3.8 [0 to 6]

2. Primary Outcome: Study Retention Rate
Description: Number of participants completing the study every 3 months.
Time Frame: From date of enrollment until either completion of study or lost to follow up every 3 months up to 2 years and 3 months
Measure: Mean (Full Range); unit: participants/3 months
Groups:
- Fluoxetine: Subjects randomized to receive fluoxetine.
- Placebo: Subjects randomized to receive placebo.
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 11 | 11
participants/3 months | 1.2 [0 to 4] | 1.1 [0 to 3]

3. Secondary Outcome: Change in Minute Ventilation During Hypercapnic Ventilatory Response (HCVR) Testing
Description: Minute ventilation was evaluated at baseline HCVR testing and HCVR testing at 4 weeks after receiving an intervention. Change from baseline was calculated.
Time Frame: At the end of HCVR testing- at baseline and 4 weeks after receiving an intervention
Population: Minute ventilation at the end of HCVR- 4 weeks after receiving an intervention was compared to minute ventilation during baseline HCVR testing in each group.
Measure: Mean (95% Confidence Interval); unit: Liters/minute (L/min)
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 11 | 11
Liters/minute (L/min) | 1.739 [-2.991 to 6.469] | 2.758 [-2.955 to 8.470]

4. Secondary Outcome: Change in PHQ-9 Score.
Description: Patient Health Questionnaire (PHQ-9) was used to evaluate mood. Score on PHQ-9 scale ranges from 0-27. Scores corresponding to severity of depression: 0-4: minimal to none ; 5-9: mild; 10-14: moderate; 15-19 moderately severe; 20-27: severe. All subjects in the study were interviewed using standard questions per PHQ-09 questionnaire at baseline and 4 weeks after randomization to an intervention.
Time Frame: At baseline and 4 weeks after randomization to an intervention
Population: PHQ-9 scores 4 weeks of receiving an intervention is compared to the baseline scores in each group.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 11 | 11
score on a scale | 0.455 [-4.309 to 5.218] | -1.000 [-4.194 to 2.194]

5. Secondary Outcome: Change in Slope of HCVR
Description: All the subjects undergo CO2 rebreathing (HCVR) testing at baseline and 4 weeks after receiving an intervention. During CO2 rebreathing (HCVR) testing, CO2 gradually rise in the body that stimulates breathing, which in turn increases minute ventilation (L/min). The rate of this increase in minute ventilation with each mm Hg rise in CO2 is the HCVR slope, which is calculated for baseline testing and 4 weeks after receiving an intervention. HCVR slope at 4 weeks after receiving an intervention compared to the baseline HCVR slope in each group.
Time Frame: At baseline and 4 weeks after receiving an intervention
Population: During CO2 rebreathing (HCVR) testing, CO2 gradually rise in the body that stimulates breathing, which in turn increases minute ventilation (L/min). The rate of this increase in minute ventilation with each mm Hg rise in CO2 is the HCVR slope, hence expressed as L/min/mm Hg unit.
Measure: Mean (95% Confidence Interval); unit: Liters/minute/mm Hg (L/min/mm Hg)
Groups:
- Fluoxetine: Subjects randomized to fluoxetine.
Arm/Group | Fluoxetine | Placebo
Number analyzed (Participants) | 11 | 11
Liters/minute/mm Hg (L/min/mm Hg) | -0.049 [-0.511 to 0.412] | 0.072 [-0.686 to 0.830]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored and collected after randomization up to 7 weeks from study drug initiation or study dropout which ever was closer.
Description: We used definition of adverse events similar to clinicaltrials.gov.
Groups:
- Fluoxetine: Subjects randomized to treatment arm will receive fluoxetine with titration schedule consisting of 10 mg per day for 1 week, 20 mg per day for 1 week, 40 mg per day for 2 weeks, 20 mg per day for 1 week and 10 mg per day for 1 week. Then stop.
  Fluoxetine: Standard 6 weeks titration, starting 10 mg per day.
- Placebo: Subjects randomized to control arm will receive placebo with titration schedule consisting of 10 mg per day for 1 week, 20 mg per day for 1 week, 40 mg per day for 2 weeks, 20 mg per day for 1 week and 10 mg per day for 1 week. Then stop.
  Placebo: Standard 6 weeks titration.
Arm/Group | Fluoxetine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 1/11 | 0/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoxetine (N=11) | Placebo (N=11)
Moderate, probably related (Nervous system disorders) | 1 (1) | 0 (0) — A subject reported feeling jittery, increased sleepiness, swollen tongue. On exam tongue was normal without any signs of swelling or other lesions. She inadvertently took higher dose than scheduled. Symptoms resolved following proper titration again.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT02929667/Prot_SAP_000.pdf